CLINICAL TRIAL: NCT06789068
Title: Lactose Intolerance in Infants With Gastrointestinal Disturbances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Haya Essam Ibrahim, lecturer of pediatrics, Ain Shams University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MS 742/ 2021
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-08

CONDITIONS: Lactose Intolerance
MeSH Terms: conditions — Lactose Intolerance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Artificially fed infants (Experimental): Infants who presented by GIT symptoms and their Cow's Milk-related Symptom Score (CoMiSS) ≥ 12 who received lactose free diet regimen for 2 weeks then received then a regimen containing lactose, a tailored dietary plan was given to each participant, and it included lactose-containing formula and dairy based products like yogurt and cheese were included for infants over 6 months.
  Interventions: Other: lactose free regimen

INTERVENTIONS:
Other: lactose free regimen — lactose free formula and solid foods that lack lactose for infants above 6 months, ensuring adequate macro and micronutrients intake according to recommended daily allowances (RDA) for age and sex.

SUMMARY:
This study enrolled thirty infants who presented by GIT symptoms and their CoMiSS was ≥ 12. The patients were assessed upon presentation, after 2 weeks of receiving lactose free diet regimen and 2 weeks after rechallenging them with lactose. Assessments of infants included anthropometric measurements, CoMiSS estimation, Neonatal/Infant Pain Scale (NIPS) and pediatric quality of life assessment (Peds QL). The study aims to detect the frequency of infants with LI with positive Cow's Milk-related Symptom Score (CoMiSS) (which could lead to misdiagnosis as CMPA) and validate of this score to be used as a screening tool for LI in infants.

ELIGIBILITY:
Inclusion Criteria:

* Artificially fed infants.
* Presented with GIT symptoms such as vomiting, diarrhea, abdominal pain, discomfort and distention.
* Cow's Milk-related Symptom Score (CoMiSS) of 12 or higher.

Exclusion Criteria:

* Infants with positive family history of Cow's milk protein allergy CMPA.
* Any allergic diseases.
* History of anaphylaxis.
* Atopic dermatitis, swelling of lips or eyelids, urticaria or wheezy chest.

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-04-13 (Actual)

PRIMARY OUTCOMES:
Frequency of infants with LI and mis diagnosed as a cow milk protein allergy. | 4 weeks intervention
  Number of infants with LI with positive Cow's Milk-related Symptom Score (CoMiSS) (which could lead to misdiagnosis as CMPA)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided